CLINICAL TRIAL: NCT01542931
Title: Study of TPF (Docetaxel, Cisplatin, 5-fluorouracil) Induction Chemotherapy Followed by Surgery and Radiotherapy in Patients With Locally Advanced and Resectable Oral Squamous Cell Carcinoma
Brief Title: TPF Induction Chemotherapy for Locally Advanced and Resectable Oral Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai-ping Zhong, Ninth People's Hospital, School of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPF for resectable OSCC; 2007BAI18B03 (Other Grant/Funding Number: National Key Technology R&D Program of China/2007BAI18B03)
Record Dates: First submitted 2012-02-26; First posted 2012-03-02 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2012-02

CONDITIONS: Stage III Oral Cavity Squamous Cell Carcinoma; Stage IVA Oral Cavity Squamous Cell Carcinoma
Keywords: Oral squamous cell carcinoma; Induction chemotherapy; Surgery; Radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery and radiotherapy (No Intervention): Surgery and post-operative radiotherapy.
- TPF induction chemotherapy (Experimental): Induction chemotherapy before surgery: docetaxel, cisplatin, and 5-fluorouracil.
  Interventions: Drug: TPF induction chemotherapy

INTERVENTIONS:
Drug: TPF induction chemotherapy — Docetaxel (at a dose of 75mg/m2 of body surface area) was administered as a 2-hour intravenous infusion, followed by intravenous cisplatin (75 mg/m2), administered during a period of 2 to 3 hours. After completion of the cisplatin infusion, 5-Fu (750 mg/m2/day) was administered during a period at least 8 hours for 5 days. Induction chemotherapy was given every 3 weeks for 2 cycles, unless there was disease progression, unacceptable toxic effects, or withdrawal of consent by the patient.
  Other Names: Followed by surgery and radiotherapy.
  Arms: TPF induction chemotherapy

SUMMARY:
Induction chemotherapy is regarded as an effective way to reduce or downgrade the locally advanced or aggressive cancers, and to improve the chance of eradication of the locoregional lesions by radical surgery and/or radiotherapy. However, there are still debates on the clinical value of induction chemotherapy for patients with advanced and resectable oral squamous cell carcinoma. The hypothesis of this study is that the induction chemotherapy of TPF (docetaxel, cisplatin, and 5-fluorouracil) protocol could benefit the patients with locally advanced oral squamous cell carcinoma. The endpoints of this study are the survival rate, local control, and safety.

DETAILED DESCRIPTION:
The primary endpoint of this study is the survival rate (2, 3, 5 years) after induction chemotherapy followed by surgery and radiotherapy. The second endpoint of this study is locoregional control rates (1, 2 years), and the safety.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study activities
* Age 18-75 years old
* Histological biopsy confirming oral squamous cell carcinoma (tongue, gingiva, buccal mucosa, floor of mouth, palate, and retromolar region)
* Clinical stage III/IVA (T1-2, N1-2, M0 or T3-4, N0-2, M0, UICC 2002), resectable lesions
* Karnofsky performance status (KPS) > 60
* Adequate hematologic function: white blood cell > 3,000/mm^3, hemoglobin > 8g/L, platelet count > 80,000/mm^3
* Hepatic function: ALAT/ASAT < 2.5 times the upper limit of normal (ULN), bilirubin < 1.5 times ULN
* Renal function: serum creatinine < 1.5 x ULN
* Life expectancy ≥ 6 months

Exclusion Criteria:

* Evidence of distant metastatic disease and other cancers
* Surgical procedure of the primary tumor or lymph nodes (except diagnostic biopsy) before study treatment
* Previous radiotherapy for the primary tumor or lymph nodes
* Prior chemotherapy or immunotherapy for the primary tumor
* Other previous malignancy within 5 years
* Systematic diseases history of severe pulmonary or cardiac diseases
* Creatinine Clearance < 30 ml/min
* Legal incapacity or limited legal capacity
* Pregnancy (confirmed by serum or urine β-HCG) or lactation period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2008-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Survival rate | Up to 5 years
  To evaluate the survival rate after TPF induction chemotherapy followed by surgery and radiotherapy.

SECONDARY OUTCOMES:
local control | Up to 5 yeas
  To evaluate the 1, 2, 3, 5-year local and regional control rate and distant metastasis rate after TPF indcution chemotherapy followed by surgery and radiotherapy
Number of participants with adverse events | Up to 5 years
  All adverse events, including serious adverse events, exposure of all study drugs and radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-yuan Zhang, MD, PhD, Study Chair — Department of Oral and Maxillofacial Surger, Ninth People's Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Ninth People's Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ju WT, Liu Y, Wang LZ, Li J, Ren GX, Sun J, Tu WY, Hu YJ, Ji T, Yang WJ, Li J, He Y, Wang YA, Zhang CP, Zhong LP, Zhang ZY. Phase III trial of docetaxel cisplatin 5-fluorouracil induction chemotherapy for resectable oral cancer suggests favorable pathological response as a surrogate endpoint for good therapeutic outcome. Cancer Commun (Lond). 2021 Mar;41(3):279-283. doi: 10.1002/cac2.12136. Epub 2021 Jan 20. No abstract available. PMID 33471949
- [Derived] Hu YJ, Sun WW, Zhao TC, Liu Y, Zhu DW, Wang LZ, Li J, Zhang CP, Zhang ZY, Zhong LP. Cyclin D1 overexpression enhances chemosensitivity to TPF chemotherapeutic agents via the caspase-3 pathway in oral cancer. Oncol Lett. 2020 Nov;20(5):154. doi: 10.3892/ol.2020.12015. Epub 2020 Aug 24. PMID 32934722
- [Derived] Yang CZ, Ma J, Zhu DW, Liu Y, Montgomery B, Wang LZ, Li J, Zhang ZY, Zhang CP, Zhong LP. GDF15 is a potential predictive biomarker for TPF induction chemotherapy and promotes tumorigenesis and progression in oral squamous cell carcinoma. Ann Oncol. 2014 Jun;25(6):1215-22. doi: 10.1093/annonc/mdu120. Epub 2014 Mar 24. PMID 24669014
- [Derived] Zhong LP, Zhang CP, Ren GX, Guo W, William WN Jr, Sun J, Zhu HG, Tu WY, Li J, Cai YL, Wang LZ, Fan XD, Wang ZH, Hu YJ, Ji T, Yang WJ, Ye WM, Li J, He Y, Wang YA, Xu LQ, Wang BS, Kies MS, Lee JJ, Myers JN, Zhang ZY. Randomized phase III trial of induction chemotherapy with docetaxel, cisplatin, and fluorouracil followed by surgery versus up-front surgery in locally advanced resectable oral squamous cell carcinoma. J Clin Oncol. 2013 Feb 20;31(6):744-51. doi: 10.1200/JCO.2012.43.8820. Epub 2012 Nov 5. PMID 23129742